CLINICAL TRIAL: NCT03747510
Title: Prospective, Single-Center, Single Arm, Feasibility Study of the PAVmed CarpX Device for the Treatment of Carpal Tunnel Syndrome
Brief Title: PAVmed CarpX Device Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PAVmed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAVmed CarpX-01-018
Record Dates: First submitted 2018-11-08; First posted 2018-11-20 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-02

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CarpX Device (Experimental): Transverse carpal ligament release with CarpX Device
  Interventions: Device: CarpX Device

INTERVENTIONS:
Device: CarpX Device — Transverse carpal ligament release with CarpX Device

SUMMARY:
To study the safety and feasibility of the CarpX device to divide and release the transverse carpal ligament in order to provide relief for Carpal Tunnel Syndrome (CTS).

DETAILED DESCRIPTION:
This is a prospective, single center, single arm, study of the CarpX device for treatment of carpel tunnel syndrome. Patients will be followed for up to 30 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years old
* Patient is scheduled to undergo carpal tunnel release surgery
* Patient has failed to respond to conservative treatment of CTS
* CTS confirmed by strong clinical signs and positive Nerve Conduction Velocity (NCV) test
* Patient, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study mandated procedures Patient is willing and able to complete follow-up requirements

Exclusion Criteria:

* Patient has a prior or current musculoskeletal or neurologic condition that limits strength, motion, or sensation in the affected hand that is unrelated to carpal tunnel syndrome.
* Patient with stiff wrist, suspected space occupying lesions or other anatomic abnormalities of the forearm, wrist or hand or other concerns related to patient anatomy such as small wrist and/or thin skin
* Prior invasive treatment of the hand or wrist for disease processes such as De Quervain's syndrome, arthritic wrist etc. on the intended treatment side
* Previous trauma/fracture or other anatomic abnormalities of the forearm, wrist or hand on the intended treatment side
* Patient has an ipsilateral injury or other conditions affecting hand function
* Patient has acute CTS resulting from an injury (e.g., fracture)
* Patient has had previous CTR surgery on the affected hand
* Patient has severe chronic median nerve neuropathy shown by the EMG and NCS that shows denervation of the thenar muscle
* Active local or systemic infection
* Known allergy to any device component
* Known severe allergy to contrast reagent that cannot be managed with premedication
* Any significant medical condition(s) that would place patient at excessive risk for surgery such as: known bleeding disorder including thrombocytopenia (platelet count < 80,000), thrombasthenia, hemophilia or Von Willebrand's disease, unstable cardiac disease, renal failure or uncontrolled diabetes
* Patient has other medical, social or psychological problem that in the opinion of the investigator precludes them from fully participating
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Device Safety defined as freedom from Serious Adverse Events probably or definitely related to the CarpX device resulting in significant morbidity. | Through 30-day
  Freedom from Serious Adverse Events probably or definitely related to the CarpX device resulting in significant morbidity.

SECONDARY OUTCOMES:
Device Technical Success: defined as the ability of the CarpX Device to perform complete division of the transverse carpel ligament. | Through 30-day
  Defined as the ability of the CarpX Device to perform complete division of the transverse carpel ligament.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Creagh, MD, Principal Investigator — Creagh & Associates
Locations (1):
- Christchurch Hospital, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.